CLINICAL TRIAL: NCT05784142
Title: Chemotherapy and Immunotherapy Induction Followed by Hypo-radiotherapy and Immunotherapy Maintenance in Locally Advanced NSCLC
Brief Title: Chemo-immunotherapy Induction Followed by Hypo-radiotherapy in LA-NSCLC(CHIC)
Acronym: CHIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Xiangzhi Zhu, M.S, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIC
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer, Non-small Cell
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHIC single arm (Experimental): Patients who have received induction immunotherapy plus chemotherapy for 2-6 cycles and met the hypoRT criteria will be enrolled into the study.
  Interventions: Radiation: hypofractionated radiation therapy

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — * Part 1: Patients who have received induction immunotherapy plus chemotherapy for 2-6 cycles and met the hypoRT criteria will be enrolled into the study.
  * Part 2: patients will be treated with hypofractionated radiation therapy in doses up to 48-60 Gy at 4 Gy per fraction.
  * Part 3: patients with partial response or stable disease after part 2 will be eligible for immunotherapy maintenance, for up to 1 years or until disease progression or unacceptable toxicity.

SUMMARY:
For unresectable locally advanced non-small cell lung cancer (LA-NSCLC), the standard treatment at present is concurrent chemoradiation therapy (CCRT) followed by durvalumab consolidation therapy. The PACIFIC study indicated a significant benefit in progression-free survival (PFS) and overall survival (OS). Notably, the PACIFIC trial only evaluated patients who had received concurrent chemoradiotherapy. Many patients are unable to tolerate concurrent chemoradiotherapy because of a poor Eastern Cooperative Oncology Group (ECOG) performance status and a high radiation pneumonitis risk for large tumors. Sequential chemoradiotherapy is therefore widely used in clinical practice for patients who cannot tolerate. In the preimmunotherapy era, CCRT showed a significant benefit in OS compared with sequential chemoradiation therapy, with an absolute improvement of 4.5% (from 10.6% to 15.1%) at 5 years. In the immunotherapy era, neoadjuvant immunotherapy plus chemotherapy resulted in significantly longer event-free survival and a higher percentage of patients with a pathological complete response than chemotherapy alone. Therefore, it is necessary to evaluate the ability of sequential immuno-chemotherapy followed by radiotherapy in patients with unresectable LA-NSCLC.

Moreover, locoregional recurrence still remain the major causes of treatment failure in the immunotherapy era. Our previous study showed that patients with stage III NSCLC treated with hypofractionated radiation therapy(hypoRT) in doses up to 60 Gy at 4 Gy per fraction had promising survival and locoregional control rates. HypoRT may also act synergistically with immunotherapy to enhance immune responses. Thus, the investigators want to exploit the survival benefit effect of immuno-chemotherapy plus sequential hypoRT in LA-NSCLC.

Based on these premises the investigators designed a single arm, phase 2 trial to determine the efficacy and safety of combining immunotherapy in association with standard chemotherapy and subsequently with hypoRT, followed by a treatment of maintenance with only immunotherapy.

The study population includes patients with NSCLC not eligible for surgery. The trial aims to evaluate the clinical outcomes, disease control, and toxicities with this regimen.

This study will last approximately 5 years and will include approximately 55 eligible patients.

DETAILED DESCRIPTION:
The study population includes patients with NSCLC not eligible for surgery. Sample size calculation was based on the GEMSTONE301 study. It was hypothesised that the hypoRT arm would improve the median PFS by 12 months (HR=0.483). A total of 50 events were requested to detect a statistically significant difference with a type I error of 5% and a type II error of 10% in a bilateral setting. Taking into account a lost-to-follow-up rate of about 5%, we planned to enroll 55 patients.

The study consists of 3 parts:

* Part 1: Patients who have received induction immunotherapy plus chemotherapy for 2-6 cycles and met the hypoRT criteria will be enrolled into the study.
* Part 2: patients will be treated with hypofractionated radiation therapy in doses up to 48-60 Gy at 4 Gy per fraction.
* Part 3: patients with partial response or stable disease after part 2 will be eligible for immunotherapy maintenance, for up to 1 years or until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide written informed consent and understand and agree to follow the research requirements and evaluation schedule.
* Age > 18 years at time of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of > 12 weeks
* Histologically- or cytologically-documented NSCLC, in locally advanced (Stage IIB-III-v.8 IASLC), without known EGFR mutations, or ALK and ROS1 rearrangements
* Patients not eligible for surgery
* Main criteria for hypoRT:

  * Residual extranodal mass is less than 7 cm in diameter on computed tomography (CT) at the end of induction immuno-chemotherapy.
  * The longitudinal length of the PTV-esophagus overlap* is less than 3 cm（*The PTV-esophagus distance of less than 0.5 cm is considered overlapping）.
  * The transverse PTV-esophagus overlap is less than one-third of esophageal lumen cross-sectional area. If exceed one-third, the longitudinal length of the overlap must be less than 1 cm.
  * Lung dose constraint: Mean lung dose≤14Gy.
* Adequate normal organ and marrow function as defined below:

  * Haemoglobin ≥9.0 g/dL (5.59 mmol/L)
  * Absolute neutrophil count (ANC) 1.5 x 109/L (> 1500/mm3)
  * Platelet count ≥100 x 109/L (100000/mm3)
  * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal.
  * Adequate renal function defined as normal serum creatinine levels or calculated creatinine clearance (according to Cockroft-Gault or by 24 hour-urine collection).

Cockcroft-Gault formula (Cockcroft and Gault 1976):

Males: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL) Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL).

* Women of childbearing age should take the urine or serum pregnancy test, and the result of which should be negtive within ≤ 72 hours before treatment. For females, who have agreed with contraception from start of investigational drug administration to 5 months after last dose of investigational drug. For males who have agreed with contraception from start of investigational drug administration to 7 months after last dose of investigational drug.
* Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Previous radiotherapy to the thorax (prior to inclusion), including radiotherapy for breast cancer
* Mixed small cell and non-small cell lung cancer histology
* Patients with severe malnutrition, with body mass index lower than 18.5kg/m2, or PG-SGA score ≥9
* Any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, autoimmune hepatitis, pituitritis, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction); Subjects with vitiligo or who have had complete remission from childhood asthma without any intervention after adulthood may be included; Asthma requiring medical intervention with bronchodilators was not included.
* Has a previous radiotherapy, chemotherapy, hormone therapy, surgery, molecular targeted therapy or immune therapy for this malignancy or for any other past malignancy;
* Any condition requiring systemic corticosteroid therapy (prednisone with a dose higher than 10 mg / day or equivalent dose of similar drugs) or other immunosuppressants within 14 days before treatment. （Excluding the following steroid regimens：Local, ophthalmic, intra-articular, nasal and inhaled corticosteroids with minimal systemic absorption；Prophylactic short-term (≤ 7 days) use of corticosteroids (e.g., prevention of contrast media allergy) or for the treatment of non-autoimmune disorders (e.g., delayed hypersensitivity caused by exposure to allergens)
* Live vaccine injection was received in ≤ 4 weeks before treatment
* A history of immunodeficiency, including HIV infection, other acquired or congenital immunodeficiency, or a history of organ or bone marrow implantation that need immunosuppressive medications.
* There are clinical symptoms or diseases of the heart that are not well controlled, such as: 1). heart failure above grade 2 by the Criteria of NYHA; 2). unstable angina pectoris; 3). myocardial infarction occurred within 1 year; 4). Clinically meaningful supraventricular or ventricular arrhythmias require treatment or intervention;
* Has severe infections（CTCAE>2 grade）within 4 weeks before treatment; basal thoracic imaging indicating active pneumonia, or other infectious situation that need oral or intravenous antibiotic treatment (excluding Prophylactic medication for antibiotics).
* A history of interstitial lung disease, non-infectious pneumonia or uncontrolled disease, including pulmonary fibrosis, acute lung disease, etc.
* Has active pulmonary tuberculosis found by CT imaging; or has active pulmonary tuberculosis less than 1 year before inclusion; or has active pulmonary tuberculosis but without standard treatment over 1 year before inclusion;
* Uncontrolled intercurrent illness including, but not limited to,, active peptic ulcer disease or gastritis, active bleeding diatheses, ongoing or active infection, including any patient known to have evidence of acute or chronic hepatitis B (positive HBV surface antigen (HBsAg) result), hepatitis C, human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent. [Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA].
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Known allergy or hypersensitivity to radiotherapy.
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease, e.g. cervical cancer in situ
  * Superficial bladder cancer without evidence of disease
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of start of induction treatment until the date of first documented progression or death from any cause, whichever came first; up to a maximum of approximately 60 months.
  PFS was defined as the time from the date of start of induction treatment until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression). Progression was defined using RECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. PFS was calculated using the Kaplan-Meier technique.

SECONDARY OUTCOMES:
Overall Survival (OS) | From baseline until death due to any cause. up to a maximum of approximately 60 months
  OS was defined as the time from the date of start of induction treatment until death due to any cause. OS was calculated using the Kaplan-Meier technique
Locoregional recurrence (LRR) | Assessed up to a maximum of approximately 60 months
  LRR was defined as time to LRR (at the site of the primary tumor or the hilar, mediastinal, or supraclavicular lymph nodes) after radiation
Distant progression-free survival (DPFS) | Assessed up to a maximum of approximately 60 months
  DPFS was defined as time to development of distant from day 1 of induction treatment
Frequency and nature of adverse reactions (ARs) and Serious Adverse Events (SAEs) | Assessed up to 60 months.
  The assessment of safety will be mainly based on adverse reactions (ARs) and the frequency and nature of SAEs. Toxicity and safety will be evaluated during each part of the program, throughout study duration.
Proportion of patients who did not progressed and who were eligible for hypoRT | At the end of part 1 of induction chemo-immunotherapy/before part 2 (assessed up to 60 months)
  The primary objective of the study is to increase the proportion of patients eligible for hypoRT after induction with immune-chemotherapy, in comparison to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangzhi Zhu, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China